CLINICAL TRIAL: NCT01561612
Title: Breastfeeding Promotion RCT and Child Metabolic Syndrome
Brief Title: Promotion of Breastfeeding Intervention Trial
Acronym: PROBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); European Union EarlyNutrition program (Unknown); University of Bristol (Other)
Responsible Party: Principal Investigator, Emily Oken, Associate Professor, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 190250; R01HD050758 (NIH); FOOD-DT-2005-007036 (Other: European Union's project on Early Nutrition Programming: Long-term Efficacy and Safety Trials); G0600705 (Other Grant/Funding Number: UK Medical Research Council); K24HD069408 (NIH); MOP-53155 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Effect of Breastfeeding on Maternal and Child Health Outcomes
Keywords: Breastfeeding; Child Health; Obesity; Blood Pressure; Asthma; Cognitive Development; Behavior; Eczema; Lung Function; Spirometry
MeSH Terms: conditions — Breast Feeding; Obesity; Asthma; Behavior; Eczema | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Breastfeeding promotion according to World Health Organization's Baby Friendly Hospital Initiative
  Interventions: Behavioral: Breastfeeding promotion and support
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Breastfeeding promotion and support — Breastfeeding promotion and support according to the World Health Organization's Baby Friendly Hospital Initiative
  Arms: Intervention

SUMMARY:
The overall goal of the PROBIT study is to investigate the influence of a randomized breastfeeding promotion intervention designed to increase the duration and exclusivity of breastfeeding ("the breastfeeding promotion intervention") on the development of maternal and child health outcomes. The hypothesis is that randomization to the intervention will be associated with lower child adiposity, lower risk of asthma and atopy, improved lung function, and improved cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Birth at one of 34 Maternity Hospitals in Republic of Belarus
* Breastfeeding initiated at birth, with no contraindications to breastfeeding
* Apgar score >=5 at 5 minutes
* Full term gestation
* Birth weight > 2500g

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17046 (Actual)
Dates: Start 1996-06; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tract infection | 12 months of age
  Occurrence of 1 or more episodes of gastrointestinal tract infection

SECONDARY OUTCOMES:
Maternal adiposity | 6.5 and 11.5 years postpartum
Child adiposity | Throughout childhood
asthma | 6.5 and 16 years
cognition | 6.5 and 16 years
dental caries | 6.5 years
child behavior | 6.5 years
vision | 16 years
lung function | 16 years
IGF-1 | Age 11.5 years
  IGF from dried bloodspots
child height | throughout childhood
  Research measures of length/height
adiponectin | age 11.5 years
  adiponectin from dried bloodspot
Apo A1 | Child age 11.5 years
  Apo A1 in dried bloodspots
glucose | child age 11.5 years
  fingerstick glucose measured by glucometer
insulin | child age 11.5 years
  insulin measured on dried blood spots
Apo B | Child age 11.5 years
  Apo B measured in dried blood spots
Child blood pressure | throughout childhood
  Research measures of blood pressure at ages 6.5, 11.5 and 16 years
Maternal blood pressure | 11.5 years postpartum
  Research measure of maternal blood pressure
Child metabolic syndrome | Age 11.5 years
Child growth | Throughout childhood
  Growth in weight, length, weight for length, BMI, and other measures
Respiratory tract infections | to age 12 months and throughout childhood
  Number of respiratory infections, from review of medical record
Atopic Eczema | Throughout childhood
  Eczema from review of medical record, parent report,and direct examination
Atopy | Age 6.5 years
  Skinprick tests for allergy
Eating Attitudes | Age 11.5 years
  Children's Eating Attitudes Test (ChEAT) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Emily Oken, MD, Principal Investigator — Harvard Pilgrim Health Care; Richard M Martin, MD, Principal Investigator — University of Bristol
Locations (1):
- Maternal and Child Health Center, Minsk, Belarus

REFERENCES:
- [Background] Kramer MS, Chalmers B, Hodnett ED, Sevkovskaya Z, Dzikovich I, Shapiro S, Collet JP, Vanilovich I, Mezen I, Ducruet T, Shishko G, Zubovich V, Mknuik D, Gluchanina E, Dombrovsky V, Ustinovitch A, Ko T, Bogdanovich N, Ovchinikova L, Helsing E. Promotion of breastfeeding intervention trial (PROBIT): a cluster-randomized trial in the Republic of Belarus. Design, follow-up, and data validation. Adv Exp Med Biol. 2000;478:327-45. PMID 11065083
- [Background] Kramer MS, Chalmers B, Hodnett ED, Sevkovskaya Z, Dzikovich I, Shapiro S, Collet JP, Vanilovich I, Mezen I, Ducruet T, Shishko G, Zubovich V, Mknuik D, Gluchanina E, Dombrovskiy V, Ustinovitch A, Kot T, Bogdanovich N, Ovchinikova L, Helsing E; PROBIT Study Group (Promotion of Breastfeeding Intervention Trial). Promotion of Breastfeeding Intervention Trial (PROBIT): a randomized trial in the Republic of Belarus. JAMA. 2001 Jan 24-31;285(4):413-20. doi: 10.1001/jama.285.4.413. PMID 11242425
- [Background] Kramer MS, Guo T, Platt RW, Shapiro S, Collet JP, Chalmers B, Hodnett E, Sevkovskaya Z, Dzikovich I, Vanilovich I; PROBIT Study Group. Breastfeeding and infant growth: biology or bias? Pediatrics. 2002 Aug;110(2 Pt 1):343-7. doi: 10.1542/peds.110.2.343. PMID 12165588
- [Background] Kramer MS, Guo T, Platt RW, Sevkovskaya Z, Dzikovich I, Collet JP, Shapiro S, Chalmers B, Hodnett E, Vanilovich I, Mezen I, Ducruet T, Shishko G, Bogdanovich N. Infant growth and health outcomes associated with 3 compared with 6 mo of exclusive breastfeeding. Am J Clin Nutr. 2003 Aug;78(2):291-5. doi: 10.1093/ajcn/78.2.291. PMID 12885711
- [Background] Kramer MS, Guo T, Platt RW, Sevkovskaya Z, Dzikovich I, Collet JP, Shapiro S, Chalmers B, Hodnett E, Vanilovich I, Mezen I, Ducruet T, Shishko G, Bogdanovich N. Does previous infection protect against atopic eczema and recurrent wheeze in infancy? Clin Exp Allergy. 2004 May;34(5):753-6. doi: 10.1111/j.1365-2222.2004.1940.x. PMID 15144467
- [Background] Kramer MS, Kakuma R. The optimal duration of exclusive breastfeeding: a systematic review. Adv Exp Med Biol. 2004;554:63-77. doi: 10.1007/978-1-4757-4242-8_7. PMID 15384567
- [Background] Kramer MS, Vanilovich I, Matush L, Bogdanovich N, Zhang X, Shishko G, Muller-Bolla M, Platt RW. The effect of prolonged and exclusive breast-feeding on dental caries in early school-age children. New evidence from a large randomized trial. Caries Res. 2007;41(6):484-8. doi: 10.1159/000108596. Epub 2007 Sep 18. PMID 17878730
- [Background] Kramer MS, Matush L, Vanilovich I, Platt R, Bogdanovich N, Sevkovskaya Z, Dzikovich I, Shishko G, Mazer B; Promotion of Breastfeeding Intervention Trial (PROBIT) Study Group. Effect of prolonged and exclusive breast feeding on risk of allergy and asthma: cluster randomised trial. BMJ. 2007 Oct 20;335(7624):815. doi: 10.1136/bmj.39304.464016.AE. Epub 2007 Sep 11. PMID 17855282
- [Background] Kramer MS. Allergy after breast feeding. Testing hypotheses: reply. BMJ. 2007 Nov 24;335(7629):1061-2. doi: 10.1136/bmj.39395.414144.80. No abstract available. PMID 18033894
- [Background] Kramer MS, Matush L, Vanilovich I, Platt RW, Bogdanovich N, Sevkovskaya Z, Dzikovich I, Shishko G, Collet JP, Martin RM, Davey Smith G, Gillman MW, Chalmers B, Hodnett E, Shapiro S; PROBIT Study Group. Effects of prolonged and exclusive breastfeeding on child height, weight, adiposity, and blood pressure at age 6.5 y: evidence from a large randomized trial. Am J Clin Nutr. 2007 Dec;86(6):1717-21. doi: 10.1093/ajcn/86.5.1717. PMID 18065591
- [Background] Kramer MS, Fombonne E, Igumnov S, Vanilovich I, Matush L, Mironova E, Bogdanovich N, Tremblay RE, Chalmers B, Zhang X, Platt RW; Promotion of Breastfeeding Intervention Trial (PROBIT) Study Group. Effects of prolonged and exclusive breastfeeding on child behavior and maternal adjustment: evidence from a large, randomized trial. Pediatrics. 2008 Mar;121(3):e435-40. doi: 10.1542/peds.2007-1248. PMID 18310164
- [Background] Kramer MS, Matush L, Vanilovich I, Platt RW, Bogdanovich N, Sevkovskaya Z, Dzikovich I, Shishko G, Collet JP, Martin RM, Smith GD, Gillman MW, Chalmers B, Hodnett E, Shapiro S. A randomized breast-feeding promotion intervention did not reduce child obesity in Belarus. J Nutr. 2009 Feb;139(2):417S-21S. doi: 10.3945/jn.108.097675. Epub 2008 Dec 23. PMID 19106322
- [Background] Kramer MS. Methodological challenges in studying long-term effects of breast-feeding. Adv Exp Med Biol. 2009;639:121-33. doi: 10.1007/978-1-4020-8749-3_10. No abstract available. PMID 19227539
- [Background] Kramer MS, Matush L, Bogdanovich N, Dahhou M, Platt RW, Mazer B. The low prevalence of allergic disease in Eastern Europe: are risk factors consistent with the hygiene hypothesis? Clin Exp Allergy. 2009 May;39(5):708-16. doi: 10.1111/j.1365-2222.2009.03205.x. Epub 2009 Mar 3. PMID 19302257
- [Background] Kramer MS, Martin RM, Sterne JA, Shapiro S, Dahhou M, Platt RW. The double jeopardy of clustered measurement and cluster randomisation. BMJ. 2009 Aug 21;339:b2900. doi: 10.1136/bmj.b2900. PMID 19700507
- [Background] Kramer MS, Matush L, Bogdanovich N, Aboud F, Mazer B, Fombonne E, Collet JP, Hodnett E, Mironova E, Igumnov S, Chalmers B, Dahhou M, Platt RW. Health and development outcomes in 6.5-y-old children breastfed exclusively for 3 or 6 mo. Am J Clin Nutr. 2009 Oct;90(4):1070-4. doi: 10.3945/ajcn.2009.28021. Epub 2009 Aug 26. PMID 19710187
- [Background] Yang S, Platt RW, Kramer MS. Variation in child cognitive ability by week of gestation among healthy term births. Am J Epidemiol. 2010 Feb 15;171(4):399-406. doi: 10.1093/aje/kwp413. Epub 2010 Jan 15. PMID 20080810
- [Background] Kramer MS. Breastfeeding, complementary (solid) foods, and long-term risk of obesity. Am J Clin Nutr. 2010 Mar;91(3):500-1. doi: 10.3945/ajcn.2010.29199. Epub 2010 Jan 27. No abstract available. PMID 20107200
- [Background] Kramer MS. Long-term behavioral consequences of infant feeding: the limits of observational studies. J Pediatr. 2010 Apr;156(4):523-4. doi: 10.1016/j.jpeds.2009.12.002. Epub 2010 Feb 10. No abstract available. PMID 20149388
- [Background] Kramer MS. "Breast is best": The evidence. Early Hum Dev. 2010 Nov;86(11):729-32. doi: 10.1016/j.earlhumdev.2010.08.005. Epub 2010 Sep 16. PMID 20846797
- [Background] Martin RM, Kramer MS, Dahhou M, Platt RW, Patel R, Bogdanovich N, Matush L, Davey Smith G; Promotion of Breastfeeding Intervention Trial (PROBIT) Study Group. Do gastrointestinal tract infections in infancy increase blood pressure in childhood? A cohort study. J Epidemiol Community Health. 2010 Dec;64(12):1068-73. doi: 10.1136/jech.2009.090894. Epub 2009 Nov 5. PMID 19897470
- [Background] Patel R, Martin RM, Kramer MS, Oken E, Bogdanovich N, Matush L, Smith GD, Lawlor DA. Familial associations of adiposity: findings from a cross-sectional study of 12,181 parental-offspring trios from Belarus. PLoS One. 2011 Jan 27;6(1):e14607. doi: 10.1371/journal.pone.0014607. PMID 21298034
- [Background] Patel R, Lawlor DA, Kramer MS, Smith GD, Bogdanovich N, Matush L, Martin RM. Socio-economic position and adiposity among children and their parents in the Republic of Belarus. Eur J Public Health. 2011 Apr;21(2):158-65. doi: 10.1093/eurpub/ckq041. Epub 2010 Apr 23. PMID 20418336
- [Background] Kramer MS, Moodie EE, Dahhou M, Platt RW. Breastfeeding and infant size: evidence of reverse causality. Am J Epidemiol. 2011 May 1;173(9):978-83. doi: 10.1093/aje/kwq495. Epub 2011 Mar 23. PMID 21430194
- [Background] Yang S, Fombonne E, Kramer MS. Duration of gestation, size at birth and later childhood behaviour. Paediatr Perinat Epidemiol. 2011 Jul;25(4):377-87. doi: 10.1111/j.1365-3016.2011.01193.x. Epub 2011 Apr 26. PMID 21649680
- [Background] Patel R, Lawlor DA, Kramer MS, Davey Smith G, Bogdanovich N, Matush L, Martin RM. Socioeconomic inequalities in height, leg length and trunk length among children aged 6.5 years and their parents from the Republic of Belarus: evidence from the Promotion of Breastfeeding Intervention Trial (PROBIT). Ann Hum Biol. 2011 Sep;38(5):592-602. doi: 10.3109/03014460.2011.577752. Epub 2011 May 19. PMID 21591995
- [Background] Tilling K, Davies N, Windmeijer F, Kramer MS, Bogdanovich N, Matush L, Patel R, Smith GD, Ben-Shlomo Y, Martin RM; Promotion of Breastfeeding Intervention Trial (PROBIT) study group. Is infant weight associated with childhood blood pressure? Analysis of the Promotion of Breastfeeding Intervention Trial (PROBIT) cohort. Int J Epidemiol. 2011 Oct;40(5):1227-37. doi: 10.1093/ije/dyr119. Epub 2011 Sep 3. PMID 22039193
- [Background] Yang S, Tilling K, Martin R, Davies N, Ben-Shlomo Y, Kramer MS. Pre-natal and post-natal growth trajectories and childhood cognitive ability and mental health. Int J Epidemiol. 2011 Oct;40(5):1215-26. doi: 10.1093/ije/dyr094. Epub 2011 Jul 15. PMID 21764769
- [Background] Kramer MS, Fombonne E, Matush L, Bogdanovich N, Dahhou M, Platt RW. Long-term behavioural consequences of infant feeding: the limits of observational studies. Paediatr Perinat Epidemiol. 2011 Nov;25(6):500-6. doi: 10.1111/j.1365-3016.2011.01211.x. Epub 2011 Jun 26. PMID 21980939
- [Background] Tilling K, Davies NM, Nicoli E, Ben-Shlomo Y, Kramer MS, Patel R, Oken E, Martin RM. Associations of growth trajectories in infancy and early childhood with later childhood outcomes. Am J Clin Nutr. 2011 Dec;94(6 Suppl):1808S-1813S. doi: 10.3945/ajcn.110.001644. Epub 2011 Jun 1. PMID 21633072
- [Background] Kramer MS. Breastfeeding and allergy: the evidence. Ann Nutr Metab. 2011;59 Suppl 1:20-6. doi: 10.1159/000334148. Epub 2011 Dec 21. PMID 22189253
- [Background] Yang S, Kramer MS. Paternal alcohol consumption, family transition and child development in a former Soviet country. Int J Epidemiol. 2012 Aug;41(4):1086-96. doi: 10.1093/ije/dys071. Epub 2012 May 13. PMID 22586132
- [Background] Kramer MS, Moodie EE, Platt RW. Infant feeding and growth: can we answer the causal question? Epidemiology. 2012 Nov;23(6):790-4. doi: 10.1097/EDE.0b013e31826cc0e9. No abstract available. PMID 23038108
- [Background] Martin RM, Patel R, Zinovik A, Kramer MS, Oken E, Vilchuck K, Bogdanovich N, Sergeichick N, Gunnarsson R, Grufman L, Foo Y, Gusina N. Filter paper blood spot enzyme linked immunoassay for insulin and application in the evaluation of determinants of child insulin resistance. PLoS One. 2012;7(10):e46752. doi: 10.1371/journal.pone.0046752. Epub 2012 Oct 8. PMID 23056434
- [Background] Patel R, Oken E, Bogdanovich N, Matush L, Sevkovskaya Z, Chalmers B, Hodnett ED, Vilchuck K, Kramer MS, Martin RM. Cohort profile: The promotion of breastfeeding intervention trial (PROBIT). Int J Epidemiol. 2014 Jun;43(3):679-90. doi: 10.1093/ije/dyt003. Epub 2013 Mar 7. PMID 23471837
- [Background] Martin RM, Patel R, Kramer MS, Guthrie L, Vilchuck K, Bogdanovich N, Sergeichick N, Gusina N, Foo Y, Palmer T, Rifas-Shiman SL, Gillman MW, Smith GD, Oken E. Effects of promoting longer-term and exclusive breastfeeding on adiposity and insulin-like growth factor-I at age 11.5 years: a randomized trial. JAMA. 2013 Mar 13;309(10):1005-13. doi: 10.1001/jama.2013.167. PMID 23483175
- [Background] Anderson EL, Fraser A, Martin RM, Kramer MS, Oken E, Patel R, Tilling K; PROBIT Study. Associations of postnatal growth with asthma and atopy: the PROBIT Study. Pediatr Allergy Immunol. 2013 Mar;24(2):122-30. doi: 10.1111/pai.12049. Epub 2013 Feb 3. PMID 23374010
- [Derived] Owen CG, Oken E, Rudnicka AR, Patel R, Thompson J, Rifas-Shiman SL, Vilchuck K, Bogdanovich N, Hameza M, Kramer MS, Martin RM. The Effect of Longer-Term and Exclusive Breastfeeding Promotion on Visual Outcome in Adolescence. Invest Ophthalmol Vis Sci. 2018 Jun 1;59(7):2670-2678. doi: 10.1167/iovs.17-23211. PMID 29860453
- [Derived] Yang S, Martin RM, Oken E, Hameza M, Doniger G, Amit S, Patel R, Thompson J, Rifas-Shiman SL, Vilchuck K, Bogdanovich N, Kramer MS. Breastfeeding during infancy and neurocognitive function in adolescence: 16-year follow-up of the PROBIT cluster-randomized trial. PLoS Med. 2018 Apr 20;15(4):e1002554. doi: 10.1371/journal.pmed.1002554. eCollection 2018 Apr. PMID 29677187
- [Derived] Flohr C, Henderson AJ, Kramer MS, Patel R, Thompson J, Rifas-Shiman SL, Yang S, Vilchuck K, Bogdanovich N, Hameza M, Martin RM, Oken E. Effect of an Intervention to Promote Breastfeeding on Asthma, Lung Function, and Atopic Eczema at Age 16 Years: Follow-up of the PROBIT Randomized Trial. JAMA Pediatr. 2018 Jan 2;172(1):e174064. doi: 10.1001/jamapediatrics.2017.4064. Epub 2018 Jan 2. PMID 29131887
- [Derived] Martin RM, Kramer MS, Patel R, Rifas-Shiman SL, Thompson J, Yang S, Vilchuck K, Bogdanovich N, Hameza M, Tilling K, Oken E. Effects of Promoting Long-term, Exclusive Breastfeeding on Adolescent Adiposity, Blood Pressure, and Growth Trajectories: A Secondary Analysis of a Randomized Clinical Trial. JAMA Pediatr. 2017 Jul 3;171(7):e170698. doi: 10.1001/jamapediatrics.2017.0698. Epub 2017 Jul 3. PMID 28459932
- [Derived] Wade KH, Kramer MS, Oken E, Timpson NJ, Skugarevsky O, Patel R, Bogdanovich N, Vilchuck K, Davey Smith G, Thompson J, Martin RM. Prospective associations between problematic eating attitudes in midchildhood and the future onset of adolescent obesity and high blood pressure. Am J Clin Nutr. 2017 Feb;105(2):306-312. doi: 10.3945/ajcn.116.141697. Epub 2016 Dec 14. PMID 27974308
- [Derived] Patel R, Tilling K, Lawlor DA, Howe LD, Bogdanovich N, Matush L, Nicoli E, Kramer MS, Martin RM. Socioeconomic differences in childhood length/height trajectories in a middle-income country: a cohort study. BMC Public Health. 2014 Sep 8;14:932. doi: 10.1186/1471-2458-14-932. PMID 25200513
- [Derived] Martin RM, Patel R, Kramer MS, Vilchuck K, Bogdanovich N, Sergeichick N, Gusina N, Foo Y, Palmer T, Thompson J, Gillman MW, Smith GD, Oken E. Effects of promoting longer-term and exclusive breastfeeding on cardiometabolic risk factors at age 11.5 years: a cluster-randomized, controlled trial. Circulation. 2014 Jan 21;129(3):321-9. doi: 10.1161/CIRCULATIONAHA.113.005160. Epub 2013 Dec 3. PMID 24300437
- [Derived] Oken E, Patel R, Guthrie LB, Vilchuck K, Bogdanovich N, Sergeichick N, Palmer TM, Kramer MS, Martin RM. Effects of an intervention to promote breastfeeding on maternal adiposity and blood pressure at 11.5 y postpartum: results from the Promotion of Breastfeeding Intervention Trial, a cluster-randomized controlled trial. Am J Clin Nutr. 2013 Oct;98(4):1048-56. doi: 10.3945/ajcn.113.065300. Epub 2013 Aug 14. PMID 23945719
- See also: Related Info — http://www.bris.ac.uk/social-community-medicine/people/project/1411